CLINICAL TRIAL: NCT01298128
Title: A Randomized Controlled Trial of NuvaRing® Versus Combined Oral Contraceptive Pills for Pre-treatment in In-Vitro Fertilization (IVF) Cycles
Brief Title: NuvaRing vs. Oral Contraceptive Pills (OCP) for In-Vitro Fertilization (IVF) Pre-treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Kimberly Liu, Physician, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFRH- 001
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Infertility; In-vitro Fertilization
MeSH Terms: conditions — Infertility | interventions — NuvaRing; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NuvaRing (Experimental): NuvaRing for IVF pre-treatment
  Interventions: Drug: NuvaRing
- Combined oral contraceptive pill (Active Comparator): OCP for IVF pre-treatment
  Interventions: Drug: marvelon

INTERVENTIONS:
Drug: NuvaRing — NuvaRIng 21 days for IVF pre-treatment.
  Arms: NuvaRing
Drug: marvelon — marvelon 21 daily
  Arms: Combined oral contraceptive pill

SUMMARY:
The newly designed contraceptive ring, Nuvaring has a lower total steroid dose, and medications are delivered locally. It has been proven to be as safe and effective as the combined OCP in ovarian suppression and preventing ovulation with fewer side effects due to minimal systemic absorption. Following a single vaginal insertion, steroid concentrations remain stable for up to 4 weeks. It is hypothesized that Nuvaring may, therefore lead to better compliance, tolerability and acceptance by patients requiring ovarian suppression prior to COH for IVF.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 38 years of age.
* Healthy women starting their first IVF/ICSI cycle.
* No contraindication to Combined Oral Contraceptive (COC) use. Appendix 1
* Consent to randomization.

Exclusion Criteria:

* Any contraindication to COC use.
* Hypersensitivity to Nuva ring or any of its components.
* Language barrier to consent.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2006-02; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly E Liu, MD, Principal Investigator — Mount Sinai Hospital, Toronto ON

REFERENCES:
- [Derived] Liu KE, Alhajri M, Greenblatt E. A randomized controlled trial of NuvaRing versus combined oral contraceptive pills for pretreatment in in vitro fertilization cycles. Fertil Steril. 2011 Sep;96(3):605-8. doi: 10.1016/j.fertnstert.2011.06.073. PMID 21880278

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NuvaRing | Combined Oral Contraceptive Pill
Started | 35 | 35
Completed | 26 | 27
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NuvaRing | Combined Oral Contraceptive Pill | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.6 (2) | 32.8 (2) | 33 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Side Effects of Oral Contraceptives Such as Abnormal Bleeding, Headache, Breast Discomfort, Bloating and Mood Swings (See Description)
Description: abnormal bleeding, intermittent bleeding, headache, breast discomfort, bloating, mood swings, nausea, vaginal discharge, vomitting, weight gain
Time Frame: patients were followed for the duration of an in-vitro fertilization cycle- 2 months
Population: 70 patients were recruited and randomized. 53 patients completed the study. 11 patients did not then undergo an ivf cycle after recruitment. 6 patients withdrew from the study after recruitment.
Measure: Number; unit: participants
Arm/Group | NuvaRing | Combined Oral Contraceptive Pill
Number analyzed (Participants) | 26 | 27
participants | 3 | 4

ADVERSE EVENTS:
Arm/Group | NuvaRing | Combined Oral Contraceptive Pill
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
early termination due to poor recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No